CLINICAL TRIAL: NCT07347106
Title: A Prospective, Randomized Controlled Trial of Miro3D Wound Matrix With Standard of Care Versus Standard of Care Alone in Treating Acute Soft Tissue Wounds and Chronic Pressure Ulcerations
Brief Title: Miro3D Randomized Controlled Trial (RCT)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202506105
Record Dates: First submitted 2025-08-19; First posted 2026-01-16 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Wound
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Intervention Model Description: Subjects will be randomly assigned to receive one of the 2 study treatments: either standard of care alone or standard of care treatment with Miro 3D. Efficacy will be determined by quantifying wound closure and PAR toward closure. The trial will also examine cost of care, number of serial placements of Miro3D, and time to hospital discharge for acute wounds.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Complex soft tissue wound arm (Active Comparator): The complex soft tissue wound arm will include consented subjects who have three-dimensional tissue defects, either elevated calf intra-compartmental hypertension treated with fasciotomy or serious infections of the foot or lower extremity that have been controlled with surgical debridement. Subjects will be randomized to either SOC alone or SOC plus Miro3D.
  Interventions: Other: Standard of Care Treatment or Standard of Care Treatment plus Miro3D Wound Matrix
- Chronic pressure ulceration arm (Active Comparator): The chronic pressure ulceration arm will include consented subjects with three-dimensional tissue deficits resulting from Stage III or greater pressure ulcerations, either a decubitus or ischial pressure ulcer that has been present and treated with SOC for at least four (4) weeks. Subjects will be randomized to SOC plus Miro3D or SOC alone.
  Interventions: Other: Standard of Care Treatment or Standard of Care Treatment plus Miro3D Wound Matrix

INTERVENTIONS:
Other: Standard of Care Treatment or Standard of Care Treatment plus Miro3D Wound Matrix — Subjects with lower extremity three-dimensional tissue defects, including those resulting from elevated calf intra-compartmental hypertension treated with decompressive fasciotomies or serious NSSTIs of the foot or lower extremities (including the pelvis as part of the lower extremity). These defects must have been controlled with surgical debridement. Subjects will be randomized to either SOC alone or SOC plus the application of Miro3D tissue scaffolding.
  Arms: Complex soft tissue wound arm
Other: Standard of Care Treatment or Standard of Care Treatment plus Miro3D Wound Matrix — Subjects with complex pressure ulcerations, particularly decubitus or ischial pressure ulcerations (Stage III or greater). These subjects will be randomized to either SOC alone or SOC plus Miro3D tissue scaffolding.
  Arms: Chronic pressure ulceration arm

SUMMARY:
The purpose of this research study is to evaluate the outcomes for patients managed with standard of care (SOC) wound treatments and those managed with standard of care treatment and tissue scaffolds, specifically Miro 3D. Tissue scaffolds like Miro 3D are 3-dimentional frameworks for collagen protein that provide structure and protection to help wounds heal.

DETAILED DESCRIPTION:
Acellular tissue scaffolds, such as Miro3D, were developed to aid in the management of complex tissue defect wounds and ulcerations by providing a structural matrix that supports cellular infiltration and tissue regeneration. However, high-quality prospective data remain limited, particularly regarding soft tissue deficits and pressure ulcerations. This prospective RCT is designed to evaluate the efficacy and outcomes of subjects randomized to receive either SOC alone or SOC with the addition of tissue scaffolding techniques (Miro3D) over a twelve (12)-week timeframe.

The trial will investigate two categories of complex wounds: soft tissue wounds, including post-fasciotomy wounds and wounds resulting from necrotizing skin and soft tissue infection (NSSTI), and chronic pressure ulcerations, with a focus on decubitus and ischial pressure ulcers. The trial aims to generate real-world data, including cost-effectiveness parameters, and features a crossover arm to evaluate the impact of delayed wound bed preparation and the application of tissue scaffolds.

Additionally, the trial will evaluate healing quality using digital wound photography and mathematical analysis of wound redness as a surrogate marker for granulation tissue formation. Time to hospital discharge will also be tracked for acute wounds to assess cost and resource utilization. By analyzing the effectiveness of Miro3D in combination with SOC, this trial seeks to provide meaningful insights into optimizing wound management strategies.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must fulfill all the following inclusion criteria to qualify for enrollment:

  1. Men or women 18-90 years of age at enrollment.
  2. Ability to sign consent by subject or LAR.
  3. Wounds in one of the two arms:

     * A. Soft tissue wounds with a minimum size of 1 cm x 1 cm surface area and a maximum size of 40 cm L x 20 cm W x 5 cm D, resulting from either post-fasciotomy or post-NSSTI, including the pelvis with the lower extremity. Fasciotomies must have undergone complete debridement and, in the opinion of a trial investigator, be appropriate for wound healing but not ready for primary closure at randomization.
     * B. Chronic, complex pressure ulcers classified as Stage III or higher, located in the decubitus or ischial region, that have not achieved at least a 50% reduction in ulcer area despite receiving documented SOC treatment for a minimum of four (4) weeks, with confirmed patient compliance.
  4. Subjects must agree to proper offloading and/or compression of the wound or ulcer throughout the trial.
  5. Written informed consent is required for digital photo imaging.
  6. For the Miro3D plus SOC arm, the wound or ulcer must have a clean base that is free of devitalized tissue or debris at the time of Miro3D placement.
  7. Subjects receiving NPWT at baseline are eligible for enrollment. The use of NPWT during the trial will be at the discretion of the treating provider.

Exclusion Criteria:

* Subjects who meet any of the following criteria will be excluded from trial participation:

  1. The PAR of the pressure ulcer arm has reduced by 50% or more after four (4) weeks of SOC.
  2. Wounds with active invasive infection not yet controlled in the opinion of a trial investigator.
  3. Wounds with vascular insufficiencies requiring revascularization.
  4. Trial investigator deems the subject has no meaningful wound healing potential (e.g., advanced cancer, severe malnutrition) and/or has conditions that seriously compromise the subject's ability to complete the trial or a known history of non-adherence to medical care.
  5. Undergoing chemotherapy.
  6. History of radiation to the area of the index wound or ulcer, regardless of time since last radiation treatment.
  7. Use of investigational drugs or therapies within thirty (30) days before screening.
  8. On dialysis.
  9. Sensitivity, allergy, or contraindication to Miro3D and/or NPWT or its components.
  10. Presence of third-degree burns.
  11. Index wound or ulcer exhibiting worsening ischemia or gangrene at screening.
  12. Subjects moving toward palliative or comfort care.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Rate of change defined as Percentage Area Reduction or PAR at four weeks after placement or not of the MIRO3D. | 4 weeks
  Rate of change

SECONDARY OUTCOMES:
Assess frequency of MIRO3D applications over a 12-week treatment period | 12 weeks
  Frequency of MIRO3D applications
Assess cost of care, including operating room time and time to hospital discharge for acute wounds | 12 weeks
  Cost of care (dollars as units of cost)
Assess NPWT use | 12 weeks
  Frequency of NPWT use
Assess cellular findings from tissue sampling | 12 weeks
  Prescence of bacteria or fungus, blood vessels and new healing cells on pathology
Assess antibiotic use | 12 weeks
  Frequency of antibiotic use
Assess pain | 12 weeks
  Subject-reported pain scores using Likert Scale, 0=No Pain - 10=Worst Possible Pain
Assess subject-reported ability to move to self-care | 12 weeks
  Patients will report if they are able to change their dressing on their own without anyone's assistance versus others having to assist (including if home health was able to be stopped) and when this occurred in their treatment course.

CONTACTS AND LOCATIONS:
Overall Officials: John Kirby, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fridman R, Rafat P, Van Gils CC, Horn D, Vayser D, Lambert JC Jr. Treatment of Hard-to-heal Diabetic Foot Ulcers With a Hepatic-derived Wound Matrix. Wounds. 2020 Sep;32(9):244-252. Epub 2020 Jun 21. PMID 32813669
- [Background] Doupis J, Veves A. Classification, diagnosis, and treatment of diabetic foot ulcers. Wounds. 2008 May;20(5):117-26. PMID 25942412
- [Background] International best practice guidelines: wound management in diabetic foot ulcers. Wounds Int. May 10, 2013. www.woundsinternational.com/resources/details/best-practice-guidelines-wound-management-diabetic-foot-ulcers
- [Background] Singh N, Armstrong DG, Lipsky BA. Preventing foot ulcers in patients with diabetes. JAMA. 2005 Jan 12;293(2):217-28. doi: 10.1001/jama.293.2.217. PMID 15644549
- [Background] NCD Risk Factor Collaboration (NCD-RisC). Worldwide trends in diabetes since 1980: a pooled analysis of 751 population-based studies with 4.4 million participants. Lancet. 2016 Apr 9;387(10027):1513-1530. doi: 10.1016/S0140-6736(16)00618-8. Epub 2016 Apr 6. PMID 27061677
- [Background] Cao X, Lin X, Li N, Zhao X, Zhou M, Zhao Y. Animal tissue-derived biomaterials for promoting wound healing. Mater Horiz. 2023 Aug 29;10(9):3237-3256. doi: 10.1039/d3mh00411b. PMID 37278612
- [Background] Chaudhari AA, Vig K, Baganizi DR, Sahu R, Dixit S, Dennis V, Singh SR, Pillai SR. Future Prospects for Scaffolding Methods and Biomaterials in Skin Tissue Engineering: A Review. Int J Mol Sci. 2016 Nov 25;17(12):1974. doi: 10.3390/ijms17121974. PMID 27898014
- [Background] Sharma S, Rai VK, Narang RK, Markandeywar TS. Collagen-based formulations for wound healing: A literature review. Life Sci. 2022 Feb 1;290:120096. doi: 10.1016/j.lfs.2021.120096. Epub 2021 Oct 26. PMID 34715138
- [Background] Ansari T, Southgate A, Obiri-Yeboa I, Jones LG, Greco K, Olayanju A, Mbundi L, Somasundaram M, Davidson B, Sibbons PD. Development and Characterization of a Porcine Liver Scaffold. Stem Cells Dev. 2020 Mar 1;29(5):314-326. doi: 10.1089/scd.2019.0069. Epub 2020 Feb 11. PMID 31854227
- [Background] Bertsch C, Marechal H, Gribova V, Levy B, Debry C, Lavalle P, Fath L. Biomimetic Bilayered Scaffolds for Tissue Engineering: From Current Design Strategies to Medical Applications. Adv Healthc Mater. 2023 Jul;12(17):e2203115. doi: 10.1002/adhm.202203115. Epub 2023 Mar 8. PMID 36807830